CLINICAL TRIAL: NCT03039517
Title: Post Thrombotic Syndrome Prevention Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: staffing change and lack of resources to conduct the study.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-01178
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Post Thrombotic Syndrome; Deep Vein Thrombosis
Keywords: Adaptive Compression Therapy Delivery System
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: subjects who meet the study entrance criteria will be randomly assigned into one of two groups using block randomization technique in a 1:1 ratio. The control group will receive care using elastic compression stocking and the intervention group will use the ACTitouch device. Stratified randomization will occur based on whether the DVT has iliac or non-iliac involvement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ACTitouch - ACT-Adaptive Compression Therapy (Experimental): a dual treatment pneumatic compression device offering two operational modes: sustained compression mode and intermittent compression mode. The device is applied to the lower leg (calf, ankle, and foot) and consists of an under-sock worn against the skin, a compression sleeve containing 4 inflatable chambers and a controller unit. The controller provides the airflow to inflate the chambers and monitors and adjusts the chamber pressure to maintain the intended treatment pressures.
  Interventions: Device: ACTitouch
- Standard Compression Stocking (Experimental): The control group will receive care using elastic compression stocking.
  Interventions: Device: Compression garments (stockings)

INTERVENTIONS:
Device: ACTitouch — The device is applied to the lower leg (calf, ankle, and foot) and consists of an under-sock worn against the skin, a compression sleeve containing 4 inflatable chambers and a controller unit. The controller provides the airflow to inflate the chambers and monitors and adjusts the chamber pressure to maintain the intended treatment pressures.
  Arms: ACTitouch - ACT-Adaptive Compression Therapy
Device: Compression garments (stockings) — Compression garments (stockings) now serve as the generally recommended standard of care for patients post DVT and will be utilized as the control compression method in this study. Compression garments utilized in this study will be "below the knee" style with a pressure range of 30-40 mmHg. If a patient does not have compression garments as indicated, these stockings will be provided.
  Arms: Standard Compression Stocking

SUMMARY:
This is a two arm, prospective, single center, randomized clinical trial. Subjects will be randomly assigned into one of two groups using block randomization technique in a 1:1 ratio. The control group will receive care using elastic compression stocking and the intervention group will use the ACTitouch device. Stratified randomization will occur based on whether the Deep Vein Thrombosis (DVT) has iliac or non-iliac involvement. Subjects will be followed for 2 years with clinic visits occurring at 1, 3, 6, 12, and 24 months.

DETAILED DESCRIPTION:
The purpose of this study is to determine if use of a pneumatic compression device (ACTitouch, Tactile Medical) is beneficial in improving or preventing the development of Post Thrombotic Syndrome (PTS). 84 patients who have a history of an acute proximal unilateral leg DVT diagnosed one or more months prior to enrollment, or diagnosed with a chronic proximal unilateral leg DVT at time of enrollment, on duplex or other imaging study will be randomized into two groups: the control group receiving the standard of care compression stockings and the intervention group receiving ACTitouch device.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age or older
* History of an acute proximal unilateral leg DVT diagnosed one or more months prior to enrollment, or diagnosed with a chronic proximal unilateral leg DVT at time of enrollment, on duplex or other imaging study (i.e MRV, CTV, venogram)
* Current anticoagulation therapy
* Physical ability to independently don ACTitouch or availability of help to place device

Exclusion Criteria:

* Current diagnosis of PTS or PTS symptoms
* Diagnosis of acute DVT less than 30 days prior to enrollment
* History of prior ipsilateral DVT
* Chronic venous insufficiency (CVI) with a CEAP 4 or greater and/or noted changes in the deep system during the diagnosing duplex
* Morbid Obesity (BMI > 45)
* Congestive heart failure with symptoms not controlled by medical intervention
* Pulmonary edema, active, with symptoms not controlled by medical intervention
* Peripheral artery disease (PAD) unless the patient has an ankle pressure of 60mmHg or more
* Walking disability (immobile)
* Women who are pregnant or trying to become pregnant
* Any other condition in which compression would be contraindicated as determined by the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Villalta Score | 2 Years
  The Villalta score is a disease score specific for PTS. It can be used to both diagnose and categorize the severity of the condition. It was developed in a cross-sectional study of 100 patients who were assessed 6 to 36 months after DVT.
  * PTS not present: 0 to 4
  * Mild PTS: 5 to 9
  * Moderate PTS: 10 to 14
  * Severe PTS: >15

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Maldonado, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States